CLINICAL TRIAL: NCT05210491
Title: The Effect of Varying Brightness Levels on Palpebral Aperture and the Point of Orbicularis Engagement Using EEG Signalling.
Brief Title: The Effect of Varying Brightness on Palpebral Aperture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Edinburgh (Other)
Collaborators: National Health Service, United Kingdom (Other Government); Royal Free Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1062/RD
Record Dates: First submitted 2022-01-14; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Eyelid Ptoses
Keywords: Palpebral Aperture measurements
MeSH Terms: conditions — Blepharoptosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The observation of eyelid positioning and EEG pulses from the eyelid on increasing brightness (Experimental): In a dimly lit room the participant will place their chin on the slit lamp We will use t he optimal background illumination used for Humphrey and Goldman visual fields which is 31.5 apostilbs (10Lux 9 They will look into the video camera placed 50cm away, which will have a dimmable remote control ring light fitted around it. The part icipant will have a reference measure taped to the headrest and three electrodes placed around the right eye. One active electrode place on the lower lid and one reference electrode towards the temporal margin and one earth electrode placed on the forehead The brightness of the ring light will be increased via the dimmer switch whilst simultaneously recording the lux with the LED light meter. The participant will be advised t o close their eyes if the brightness becomes uncomfortable and this will be repea ted three times.
  Interventions: Other: Review of eyelid positioning in increasing brightness levels

INTERVENTIONS:
Other: Review of eyelid positioning in increasing brightness levels — Up to 30 seconds, three times, looking into a video camera as glare is incrementally increased.

SUMMARY:
We aim to establish the point at which glare from bright lights begins to engage our eyelids - causing us to "squint". We will be using a video camera with an LED ring light around it facing the volunteer and we will record the eyelid position as the light brightness is increased gradually. Many studies have looked at the effect glare has on a person through qualitative questionnaires but few have been able to quantify this.

DETAILED DESCRIPTION:
Our study will aim to establish the point of orbicularis engagement based on luminous intensity Murray et al. created an Ocular Stress Monitor to see if the contracture of the muscles on the eyelid indicative of pain as a light source was increased in luminosity 8 Our study will go one step further by using video technology and a portable EEG machine to detect the pulses of lid contracture as luminosity of a ring light i s increased incrementally. An advanced calibrated datalogging LED light meter will simultaneously record the level of brightness to establish at which point the spike in EEG occurs. Screenshots from the video recording will be taken and accurate MRD1 measurements can be taken at the point of orbicular i s engagement.

The scientific justification for this research question is twofold We wish to establish the threshold at which orbicularis engages such that palpebral aperture and MRD measurements are altered. This is relevant to the technique of taking these measurements in the clinical environment and the light intensity at which these measurements are taken. We wish to establish the light intensity which should not be exceeded to take these measurements. As photography becomes increasingly used in oculoplastic s clinics we envisage palpebral aperture and MRD1 measurements being performed digitally rather than manually These measurements are relevant to pre operative and post operative imaging, and surgical planning. Furthermore, our results maybe applicable more widely to industry, for example vehicle headlights, bicycle lights, camera flash, workplace lighting.

Reference: Murray I, Plainis S, Carden D. The ocular stress monitor: a new device for measuring discomfort glare. Lighting Research Technology. 2002;34(3):231 239.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years of age
* A member of the Royal Free NHS trust

Exclusion Criteria:

* No known ocular pathology
* No lid problems/ptosis or previous lid surgery
* No contact lenses in for duration of experiment
* No pseudophakia
* No neurological disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-14 (Actual); Primary Completion 2022-02-21 (Estimated); Study Completion 2022-02-21 (Estimated)

PRIMARY OUTCOMES:
The point at which the eyelid begins to contract under what brightness level | All carried out within a 2 week period
  Using a light meter, ring light, and EEG machine

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmology, Royal Free Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Data findings will be presented to the department, all those involved at the next departmental meeting.